CLINICAL TRIAL: NCT05210374
Title: Disulfiram With Copper Gluconate and Liposomal Doxorubicin in Patients With Treatment-Refractory Sarcomas
Brief Title: Disulfiram With Copper Gluconate and Liposomal Doxorubicin in Treatment-Refractory Sarcomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1720
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Relapsed Sarcomas
Keywords: Sarcoma,; osteosarcoma; rhabdomyosarcoma; Ewing sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Sarcoma, Ewing | interventions — Disulfiram; Gluconates; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DSF/Cu (Experimental): A 3+3 dose escalation design will be used to determine the recommended phase 2 dose (RP2D) of DSF/Cu in combination with liposomal doxorubicin. There will be a 7 day "lead-in" week of Disulfiram (DSF)/Copper Gluconate (Cu). The disulfiram and the copper gluconate will be dosed once a day. Disulfiram in the morning and copper gluconate in the evening. Same total daily dose every 4 week (28 days) administration of liposomal doxorubicin (Doxil) 30mg/m2/dose IV
  Cycle length: 28 days Maximum 12 cycles
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate; Drug: Liposomal Doxorubicin (Doxil)

INTERVENTIONS:
Drug: Disulfiram — To be taken orally (PO) daily in the AM, rounded for pill size (max 480mg/day).
  To be administered day 1-7 of lead-in week and day 1-28 cycles
  Cycle length: 28 days,
  maximum 12 cycles Level -1 (150mg/m^2/day) Level
  0 (225mg/m^2/day) Level 1 (300mg/m^2/day), max
  480mg/day
Drug: Copper Gluconate — To be taken orally (PO), 5.2mg/m2/day daily in the PM, rounded
  for pill size (max 9mg/day) To be administered day 1-7
  Lead-in week and day 1-28 cycles Cycle length: 28
  days, maximum 12 cycles
Drug: Liposomal Doxorubicin (Doxil) — To be given IV, 30mg/m2/dose
  To be administered day 1 of cycles
  Cycle length: 28 days, maximum 12 cycles
  Other Names: Pegylated Liposomal Doxorubicin (PLD); Doxorubicin HCl Liposome Injection; Dox-SL

SUMMARY:
The purpose of this study is to test the safety of combining the disulfiram (DSF) and copper gluconate (Cu) to liposomal doxorubicin to treat patients with sarcomas that recurred or did not respond to initial treatment.

DETAILED DESCRIPTION:
DSF blocks an enzyme called aldehyde dehydrogenase (ALDH). ALDH breaks down substances in the body that can be toxic. ALDH also appears to be important for making many cancers resistant to chemotherapy drugs like liposomal doxorubicin. The study team believes giving DSF with liposomal doxorubicin will help make the cancers sensitive to the liposomal doxorubicin, making it work better. Cu is an FDA approved dietary food supplement and has been shown in laboratory research to improve how DSF works, which is the rational for giving DSF with Cu. It is currently unknown if and at what dose DSF is safe to be given in this combination. Though DSF has been used for over 60 years for the treatment of alcoholism, this is the first time DSF/Cu is being tested in combination with liposomal doxorubicin in humans.

The primary objectives of this study are to:

Measure the feasibility, safety and tolerability of DSF/Cu in combination with liposomal doxorubicin

Secondary objectives of this study are to:

Measure tumor response, survival, and pharmacokinetics of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed relapsed or refractory sarcoma.
* Must have measurable disease by RECIST criteria at study enrollment
* Performance status of Karnofsky/Lansky ≥50%
* Must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine ≤1.5X institutional limit of normal
* Must be able to swallow pills or consume the contents of the DSF and Capsules sprinkled on food.
* Participants, or parent/guardians for participants <18 years old (yo), must have the ability to understand and the willingness to sign a written informed consent document.
* Must abstain from alcohol during study.
* Prior treatment toxicities must have stabilized or resolved to ≤ Grade 1 according to NCI CTCAE Version 5.0 except alopecia, neuropathy and hematologic criteria (must meet normal organ and marrow function criteria above).
* Participants ≥18yo must agree to pre-and post-treatment core needle tumor biopsies. For participants <18yo biopsies are optional. Biopsies will not be performed if deemed unsafe by interventional radiologists that will be performing the procedure and is not part of the study team to avoid bias.
* Must abstain from sexual intercourse or used appropriate, highly-effective birth control measures.

Exclusion Criteria:

* Has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Has a history of allergy or hypersensitivity to any of the study drugs, their pharmaceutical class or any of their excipients. The participant exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of Liposomal Doxorubicin Prescribing Information package inserts or on the Investigator's Brochure for DSF/Cu.
* Has a concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the participant's safety or the study data integrity.
* Is currently enrolled in any other clinical protocol or investigational trial involving administration of antineoplastic compounds for the treatment of their sarcoma.
* Is unwilling or unable to comply with study procedures.
* Know condition preventing safe administration of copper such as a copper allergy or Wilson's Disease.
* Investigator feels participation in this study would be harmful or of no benefit to the potential participant

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by percent of participants experiencing grade 3+ with at least possible attribution to study drug using CTCAE 5.0 guidelines | up to 30 days after last treatment
  Safety as measured by percent of participants experiencing grade 3+ with at least possible attribution to study drug using CTCAE 5.0 guidelines
Recommended phase 2 dose (RP2D) of DSF/Cu in combination with liposomal doxorubicin | at end of cycle 1 (day 28)
  RP2D of DSF/Cu in combination with liposomal doxorubicin
Number of participants able to take at least 80% of the drug doses during the first cycle of treatment | up to 30 days after last treatment
  Feasibility: Number of participants able to take at least 80% of the drug doses during the first cycle of treatment, assessed by the medication diary patients will be asked to keep
Number of dose-limiting toxicities (DLT) | up to 30 days after last treatment
  Tolerability, as total number of defined as number of DLTs
Number of participants who experienced drug-attributed grade 3+ Adverse events per CTCAE5.0 | up to 30 days after last treatment
  Number of participants who experienced drug-attributed grade 3+ Adverse events per CTCAE5.0

SECONDARY OUTCOMES:
Percent of participants with tumor response evaluated using RECIST v1.1 | At 2 months
  Tumor response will be evaluated per RECIST v1.1 criteria - percent of participants with complete response, partial response, stable disease and progressive disease reported
Median Overall Survival (OS) | up to 30 days after last treatment
  Median OS defined as the time from participant enrollment on study to time of death
Median Event free survival | up to 30 days after last treatment
  Median Event free survival defined as the time from participant enrollment on study to time of disease progression (PD) per RECIST v1.1,.
  PD defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [Peak concentration (Cmax)] | At hour 0 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - Peak concentration (Cmax)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [Peak concentration (Cmax)] | At hour 2 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - Peak concentration (Cmax)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [Peak concentration (Cmax)] | At hour 4 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - Peak concentration (Cmax)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [Peak concentration (Cmax)] | At hour 24 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - Peak concentration (Cmax)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [Peak concentration (Cmax)] | Day 1 of cycle 1 (day 8)
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - Peak concentration (Cmax)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [area under the concentration-vs-time curve (AUC)] | At hour 0 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - area under the concentration-vs-time curve (AUC)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [area under the concentration-vs-time curve (AUC)] | At hour 2 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - area under the concentration-vs-time curve (AUC)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [area under the concentration-vs-time curve (AUC)] | At hour 4 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - area under the concentration-vs-time curve (AUC)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [area under the concentration-vs-time curve (AUC)] | At hour 24 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - area under the concentration-vs-time curve (AUC)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [area under the concentration-vs-time curve (AUC)] | Day 1 of cycle 1 (day 8)
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - area under the concentration-vs-time curve (AUC)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [clearance and average steady state concentrations for disulfiram and its active metabolites] | At hour 0 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - clearance and average steady state concentrations for disulfiram and its active metabolites, S-methyl N,N-dietylthiolcarbamate (DETC-ME) and bis-diethyldithiocarbamate-copper complex (CuET)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [clearance and average steady state concentrations for disulfiram and its active metabolites] | At hour 2 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - clearance and average steady state concentrations for disulfiram and its active metabolites, S-methyl N,N-dietylthiolcarbamate (DETC-ME) and bis-diethyldithiocarbamate-copper complex (CuET)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [clearance and average steady state concentrations for disulfiram and its active metabolites] | At hour 4 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - clearance and average steady state concentrations for disulfiram and its active metabolites, S-methyl N,N-dietylthiolcarbamate (DETC-ME) and bis-diethyldithiocarbamate-copper complex (CuET)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [clearance and average steady state concentrations for disulfiram and its active metabolites] | At hour 24 of Day 1 of lead-in week
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - clearance and average steady state concentrations for disulfiram and its active metabolites, S-methyl N,N-dietylthiolcarbamate (DETC-ME) and bis-diethyldithiocarbamate-copper complex (CuET)
Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicin [clearance and average steady state concentrations for disulfiram and its active metabolites] | Day 1 of cycle 1 (day 8)
  Pharmacokinetics of DSF/Cu in combination with liposomal doxorubicinbased on samples collected - clearance and average steady state concentrations for disulfiram and its active metabolites, S-methyl N,N-dietylthiolcarbamate (DETC-ME) and bis-diethyldithiocarbamate-copper complex (CuET)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Trucco, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and for 3 years following publication
Access Criteria: Researchers who provide a sound rationale for access